CLINICAL TRIAL: NCT00819936
Title: A Controlled Trial of Effectiveness of a Backward Walking Program in Patients Recovering From an Abdominal Aorta Surgery
Brief Title: A Controlled Trial of Effectiveness of a Backward Walking Program in Patients Recovering From Abdominal Aorta Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Medcial Univeristy of Silesia, Department of Rehabilitation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B.W 2008/A
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Abdominal Surgery
Keywords: abdominal aorta surgery; Physical Training; backward walking; physiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Backward walking,
  Interventions: Procedure: backward walking
- 1 (Active Comparator): Forward walking
  Interventions: Procedure: forward walking

INTERVENTIONS:
Procedure: forward walking — comparison forward walking vs backward walking in the physiotherapy after after abdominal surgery
  Arms: 1
Procedure: backward walking — physiotherapy with use a backward walking type of physiotherapy
  Arms: 2

SUMMARY:
Summary Question: Does backward walking offer additional therapeutic value in patients after aortic aneurysm surgery? Participants: The study of backward walking as an addictive physiotherapy procedure was conducted in the group of 65 patients who underwent abdominal aorta surgery. The patients were randomly divided into three subgroups and three various models of physiotherapy were applied. Control group has only routine physiotherapy since therapeutic group I and II have also walking exercises forward in group I and backward in group II respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abdominal aortic aneurysm
* Age 65-75 years
* Male sex
* Stable cardiologic status
* Absence of neurological disorders
* Non-symptomatic aneurysm - non-ruptured
* No pain complaints
* No motion system impairments

Exclusion Criteria:

* Patients with neurological disorders
* Unstable coronary heart disease symptomatic aortic aneurysm - dissecans aneurysm
* Having difficulty in locomotion
* Having contradiction for starting physical training during the first or second day after surgery
* Patients with psychiatric disease
* Lack of patient's compliance with physiotherapist; AND
* Other medical contraindications

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2006-12